CLINICAL TRIAL: NCT02162511
Title: An Expanded Access Study Using the CliniMACS System to Offer Therapeutic Manipulated Grafts That Are CD34 Cell Enriched and T Cell Depleted for Allogeneic Stem Cell Recipients With Mismatched Related Donors or Borderline Organ Function
Brief Title: CD34+ Cell Enriched and T Cell Depleted Allogeneic Stem Cell Transplantation for Patients With Mismatched Related Donors or Borderline Organ Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rajni Agarwal (Other)
Responsible Party: Sponsor-Investigator, Rajni Agarwal, Principal Investigator, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 28663
Record Dates: First submitted 2014-06-10; First posted 2014-06-12 (Estimated); Results first posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-05

CONDITIONS: Malignant Diseases; Non-malignant Diseases
Keywords: Haplocompatible; Stem cell transplant; Borderline organ function; Alternative donor stem cell transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- ARM A Malignant TBI (Experimental): Malignant diseases Conditioning including total body irradiation and chemotherapy
  Interventions: Device: CliniMACS CD34+ cell enrichment and T-cell depletion
- ARM B Malignant Non-TBI (Experimental): Malignant diseases chemotherapy based conditioning
  Interventions: Device: CliniMACS CD34+ cell enrichment and T-cell depletion
- ARM C Non-malignant (Experimental): Non-malignant diseases Chemotherapy based conditioning
  Interventions: Device: CliniMACS CD34+ cell enrichment and T-cell depletion

INTERVENTIONS:
Device: CliniMACS CD34+ cell enrichment and T-cell depletion

SUMMARY:
The purpose of this protocol is to provide access to the CliniMACS® System to hematopoietic cell transplant (HSCT) patients who do not have a matched related donor. The CliniMACS system is currently approved for use in patients who have AML, and a genetically matched sibling donor. Through this protocol, the investigators will be able to offer potentially life-saving transplants to patients who have genetically mis-matched donor, who have no other options for treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participant age is 0 (newborn) to 35 years-old.
* Participant has a disorder affecting the hematopoietic system that are inherited, acquired, or a result from the myeloablative treatment that can benefit from alternative stem cell transplantation according to standard practice guidelines for including patients for transplant.
* Participant's medical screening clears s/he for allogeneic transplantation as per current institutional SOP based on standards of foundation for accreditation of cellular therapy and stem cell transplantation (FACT);
* Participant must lack a healthy, HLA-identical related or unrelated donor unless s/he has a borderline organ function that will preclude the recipient from receiving a curative therapy due to the need of post-HSCT immunosuppressive therapy.
* Participant must have a matched or mismatched-related donor who is:
* Able to receive granulocyte colony-stimulating factor (G-CSF) and undergo apheresis either through placement of catheters in antecubital veins or a temporary central venous catheter OR agrees on a bone marrow harvest;
* Healthy as per donor selection screening (following current SOP based on standards of foundation for accreditation of cellular therapy and stem cell transplantation - FACT);
* Willing to participate and sign consent.
* Participant or Legal Authorized Representative is able to sign informed consent (and signed assent, if applicable) for transplant.

Exclusion Criteria:

* Participant does not qualify for an allogeneic transplant due to medical screening, underlying disease, or lack of alternative donors.
* Any condition that compromises compliance with the procedures of this protocol, as judged by the principal investigator.

Max Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2014-05; Primary Completion 2019-07 (Actual); Study Completion 2023-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajni Agarwal, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Children's Hospital, Palo Alto, California, United States

REFERENCES:
- See also: Stanford Stem Cell Transplantation website — https://med.stanford.edu/ptrm.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was open to participants with malignant or non-malignant disorders receiving mismatched related donor hematopoietic stem cell transplants who could benefit from augmented CD34+ cells and T cell-depleted products to prevent severe (grade III/IV) acute Graft vs Host Disease (GVHD). Participants were withdrawn from the study at the time of graft failure due to need for exclusionary concurrent treatment (per PI discretion)
Groups:
- ARM A Malignant TBI: Malignant diseases Conditioning including total body irradiation and chemotherapy
  CliniMACS CD34+ cell enrichment and T-cell depletion
- ARM B Malignant Non-TBI: Malignant diseases chemotherapy based conditioning
  CliniMACS CD34+ cell enrichment and T-cell depletion
- ARM C Non-malignant: Non-malignant diseases Chemotherapy based conditioning
  CliniMACS CD34+ cell enrichment and T-cell depletion
Period: Overall Study
Arm/Group | ARM A Malignant TBI | ARM B Malignant Non-TBI | ARM C Non-malignant
Started | 0 | 0 | 3
Achieved Engraftment | 0 | 0 | 1
Completed | 0 | 0 | 1
Not Completed | 0 | 0 | 2
Not completed — Lack of Efficacy | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Malignant Arms did not recruit due to other available studies for these patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | ARM A Malignant TBI | ARM B Malignant Non-TBI | ARM C Non-malignant | Total
Number analyzed (Participants) | 0 | 0 | 3 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 3 | 3
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] |  |  | 7.47 [0.4 to 17] | 7.47 [0.4 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  |  | 1 | 1
  Male |  |  | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  |  | 2 | 2
  Not Hispanic or Latino |  |  | 1 | 1
  Unknown or Not Reported |  |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  |  | 0 | 0
  Asian |  |  | 1 | 1
  Native Hawaiian or Other Pacific Islander |  |  | 0 | 0
  Black or African American |  |  | 0 | 0
  White |  |  | 0 | 0
  More than one race |  |  | 0 | 0
  Unknown or Not Reported |  |  | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States |  |  | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Severe (Grade III/IV) Acute Graft vs Host Disease (GVHD)
Description: GVHD is a condition that occurs when donor bone marrow or stem cells attack the recipient.
Time Frame: Day +100
Measure: Count of Participants; unit: Participants
Arm/Group | ARM C Non-malignant
Number analyzed (Participants) | 3
Participants | 0

2. Secondary Outcome: Number of Participants With Graft Failure
Description: Failure of donor stem cells to make neutrophils
Time Frame: Up to Day +42 after stem cell transplant
Measure: Count of Participants; unit: Participants
Arm/Group | ARM C Non-malignant
Number analyzed (Participants) | 3
Participants | 2

3. Secondary Outcome: Length of Time to Engraftment
Description: Absolute neutrophil count (ANC) >500 for 3 consecutive days and >80% donor cells in blood.
Time Frame: up to +1 year post-transplant
Population: Patients who had primary graft failure were withdrawn from the study are excluded from the analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | ARM C Non-malignant
Number analyzed (Participants) | 1
days | 10 (NA) — Standard Deviation not calculable for one participant

4. Secondary Outcome: Chimerism of Donor Cells
Description: The percentage of donor cells for all evaluable (without disease progression) patients
Time Frame: Day +100 post-transplant
Population: Patients who had primary graft failure were withdrawn from the study are excluded from the analysis.
Measure: Mean (Standard Deviation); unit: Percentage of cells from donor
Arm/Group | ARM C Non-malignant
Number analyzed (Participants) | 1
Percentage of cells from donor
  Whole Blood | 95 (NA) — Standard Deviation not calculable for one participant
  CD3 Cells | 70 (NA) — Standard Deviation not calculable for one participant
  CD15 Cells | 100 (NA) — Standard Deviation not calculable for one participant
  CD19 | 99 (NA) — Standard Deviation not calculable for one participant
  CD34 | 98 (NA) — Standard Deviation not calculable for one participant
  CD56 | 99 (NA) — Standard Deviation not calculable for one participant

5. Secondary Outcome: Immune Recovery (CD4)
Description: The time to CD4 count >100
Time Frame: up to +1 year post-transplant
Population: Patients who had primary graft failure and were withdrawn from the study are excluded from the analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | ARM C Non-malignant
Number analyzed (Participants) | 1
days | 148 (NA) — Standard Deviation not calculable for one participant

6. Secondary Outcome: Number of Participants With Immune Recovery (CD4 >200) by Year 1
Time Frame: up to +1 year post-transplant
Population: Patients who had primary graft failure and were withdrawn from the study are excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | ARM C Non-malignant
Number analyzed (Participants) | 1
Participants | 0

7. Secondary Outcome: Immune Recovery Shown as Phytohemagglutin (PHA)
Description: Immune recovery defined as achieving normal levels of PHA (53,000-200,000 CPM)
Time Frame: 6 months and 1 year post-transplant
Population: Participants who had primary graft failure were withdrawn from the study and unable to be evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: Net CPM
Arm/Group | ARM C Non-malignant
Number analyzed (Participants) | 1
Net CPM
  6 months | 33736 (NA) — Standard Deviation not calculable for one participant
  1 year | 110809 (NA) — Standard Deviation not calculable for one participant

8. Secondary Outcome: Number of Patients With Post-transplant Lymphoproliferative Disease (PTLD)
Description: Post-transplant lymphoproliferative disorder (PTLD) is a well-known, life-threatening complication of organ transplantation, predominantly occurring after solid organ transplantation (SOT) and hematopoietic stem cell transplantation (HSCT).
Time Frame: up to +1 year post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | ARM C Non-malignant
Number analyzed (Participants) | 3
Participants | 0

9. Secondary Outcome: Number of Patients With Severe Toxicities
Description: Incidence of transplant-related toxicities
Time Frame: up to +1 year post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | ARM C Non-malignant
Number analyzed (Participants) | 3
Participants | 2

10. Secondary Outcome: Number of Participants Experiencing Post-transplant Infections
Description: Post-transplant infections will be described by incidence and type. Participants may have had more than one type of infection.
Time Frame: up to +1 year post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | ARM C Non-malignant
Number analyzed (Participants) | 3
Participants
  BK viremia | 1
  BK viruria | 1
  Norovirus | 1
  HHV6 viremia | 2
  EBV viremia | 1
  Rhinovirus/Enterovirus | 1
  Parainfluenza 3 upper respiratory infection | 1
  Adenovirus (low level reactivation) | 1
  Cytomegalovirus (low level reactivation) | 1

11. Secondary Outcome: Transplant-related Mortality (TRM)
Description: Death related to transplant
Time Frame: at Day +100 and +1 year post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | ARM C Non-malignant
Number analyzed (Participants) | 3
Participants
  Day 100 | 1
  Between Day 100 and 1 Year | 1

ADVERSE EVENTS:
Time Frame: Up to 1 year post-transplant.
Description: Recipients of allogeneic hematopoietic cell transplantation face significant risks. The risk of treatment related morbidity and mortality following allogeneic transplant is related to the underlying disease, disease status at the time of transplant, prior therapies and other coexisting health problems. Therefore, in accordance with the study protocol, only AE's found to be directly related to the study-mandated intervention were captured.
Arm/Group | ARM C Non-malignant
All-Cause Mortality (participants affected / at risk) | 2/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
This study did not meet its planned enrollment. Statistical power was not achieved for any analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-02): https://cdn.clinicaltrials.gov/large-docs/11/NCT02162511/Prot_SAP_000.pdf